CLINICAL TRIAL: NCT00108277
Title: Respiratory Dysregulation and Breathing Training in Anxious Outpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHBA-028-04S
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Anxiety
Keywords: Anxiety; Breathing Training; Respiratory Dysregulation
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Raise CO2 (Experimental): Raise CO2 - biofeedback-assisted breathing training to raise baseline pCO2
  Interventions: Behavioral: Breathing Training-Raise CO2
- Lower CO2 (Active Comparator): Lower CO2 - biofeedback-assisted breathing training to lower baseline pCO2
  Interventions: Behavioral: Breathing Training- Lower CO2
- Waitlist (No Intervention): Waitlist - treatment as usual

INTERVENTIONS:
Behavioral: Breathing Training-Raise CO2 — while breathing 9 breaths per minute, patients are instructed to raise CO2
  Arms: Raise CO2
Behavioral: Breathing Training- Lower CO2 — while breathing 9 breaths per minute, patients are instructed to lower CO2
  Arms: Lower CO2

SUMMARY:
This study will explore respiratory dysregulation in anxious outpatients and examine the effect of breathing training with biofeedback for those anxious patients.

DETAILED DESCRIPTION:
In clinic testing and outside the clinic testing, we will assess the prevalence of respiratory dysregulation in a sample of 60 non-psychotic, not currently alcohol or drug abusing veteran outpatients from our MHC (Mental Hygiene Clinic) who experience episodic anxiety but who do not qualify and have never qualified for the diagnosis of PD (panic disorder). These patients will be compared to 30 patients who are not clinically anxious. Of these 60 anxious patients, 30 will be randomly assigned to a 4-week course of breathing training assisted by feedback of end-tidal pCO2 levels as an augmentation of their current treatment. They will be compared to 30 who simply will continue with their current treatment (TAU). The breathing training group will receive clinical and physiological assessments immediately before the treatment period, four weeks after the end of the treatment period, and at a 4-month follow-up. The TAU group will be assessed three times at equivalent intervals, and if they wish, may undergo breathing training after the third assessment. Treatment will take place mainly in the first two years, giving us adequate time for follow-up and data analysis. We expect that this therapy will be especially effective for treating anxiety in the patients with substantial respiratory dysregulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be rated 2 or more on both Q1 and Q3, but they must not meet the full criteria for PD as determined by the Anxiety Disorders Interview Schedule for DSM-IV-Lifetime Version (ADIS).
* In addition, they must be clinically stable enough that changes in the patients' anxiety levels can be attributed to the breathing training rather than to other new treatment initiatives during the training and 1-month evaluation periods or to spontaneous fluctuations in anxiety levels. Thus, potential participants taking SSRIs or other antidepressants, or benzodiazepines have to have been on a stable dose of these medicines for at least the previous two months.

Exclusion Criteria:

* Potential participants taking short-acting benzodiazepines such as alprazolam in excess of 2.0 mg/day or the equivalent on any day in the past month are excluded, because improvement might show up only in terms of reduction of medication dosage and not on the evaluation measures planned.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2005-04; Primary Completion 2008-12 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walton Roth, MD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Result] Wollburg E, Roth WT, Kim S. Effects of breathing training on voluntary hypo- and hyperventilation in patients with panic disorder and episodic anxiety. Appl Psychophysiol Biofeedback. 2011 Jun;36(2):81-91. doi: 10.1007/s10484-011-9150-5. PMID 21373936
- [Result] Doberenz S, Roth WT, Wollburg E, Maslowski NI, Kim S. Methodological considerations in ambulatory skin conductance monitoring. Int J Psychophysiol. 2011 May;80(2):87-95. doi: 10.1016/j.ijpsycho.2011.02.002. Epub 2011 Feb 21. PMID 21320551

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from October 2005 to September 2008 from the local VA medical center and surrounding community. Participants were primarily recruited via posted flyers and other public advertisements (e.g., ads in local newspapers).
Groups:
- Raise CO2: Raise CO2
  Breathing Training-Raise CO2: while breathing 9 minutes per minute, patients are instructed to raise CO2
- Lower CO2: Lower CO2
  Breathing Training- Lower CO2: while breathing 9 minutes per minute, patients are instructed to lower CO2
- Waitlist: Waitlist Treatment as Usual
Period: Overall Study
Arm/Group | Raise CO2 | Lower CO2 | Waitlist
Started | 29 | 28 | 35
Completed | 19 | 16 | 19
Not Completed | 10 | 12 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raise CO2 | Lower CO2 | Waitlist | Total
Number analyzed (Participants) | 29 | 28 | 35 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (13.2) | 40.6 (12.2) | 49.9 (10.9) | 45.9 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 25 | 61
  Male | 13 | 8 | 10 | 31
Race/Ethnicity, Customized [Number; unit: participants]
  White | 15 | 16 | 17 | 48
  Other | 14 | 12 | 18 | 44
Episodic Anxiety Scale [Mean (Standard Deviation); unit: units on a scale] — Episodic Anxiety Scale (EAS) is a modification of the Panic Disorder Severity Scale (Shear et al., 1997) that includes 2 additional questions regarding acute anxiety episodes that may not meet full criteria for a panic attack. The EAS consists of 9 questions, each ranging from 0 (none) to 4 (worst possible). The EAS total score is the sum of all 9 items, such that the minimum total score = 0 (no anxiety symptoms) and maximum total score = 36 (worst possible anxiety symptoms).
  units on a scale | 15.5 (3.44) | 15.7 (4.53) | 16.1 (3.23) | 15.8 (3.73)

OUTCOME MEASURES:

1. Primary Outcome: Episodic Anxiety Scale
Description: Episodic Anxiety Scale (EAS) is a modification of the Panic Disorder Severity Scale (Shear et al., 1997) that includes 2 additional questions regarding acute anxiety episodes that may not meet full criteria for a panic attack. The EAS consists of 9 questions, each ranging from 0 (none) to 4 (worst possible). The EAS total score is the sum of all 9 items, such that the minimum total score = 0 (no anxiety symptoms) and maximum total score = 36 (worst possible anxiety symptoms).
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Raise CO2: Raise CO2
  Breathing Training-Raise CO2: while breathing 9 breaths per minute, patients are instructed to raise CO2
- Lower CO2: Lower CO2
  Breathing Training- Lower CO2: while breathing 9 breaths per minute, patients are instructed to lower CO2
Arm/Group | Raise CO2 | Lower CO2 | Waitlist
Number analyzed (Participants) | 19 | 16 | 19
units on a scale | 8.1 (2.73) | 9.0 (3.89) | 14.3 (3.67)

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Raise CO2: Breathing Training-Raise CO2: while breathing 9 minutes per minute, patients are instructed to raise CO2
- Lower CO2: Breathing Training- Lower CO2: while breathing 9 minutes per minute, patients are instructed to lower CO2
- Waitlist: Treatment as usual
Arm/Group | Raise CO2 | Lower CO2 | Waitlist
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28 | 0/35
Other Adverse Events (participants affected / at risk) | 0/29 | 0/28 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No